CLINICAL TRIAL: NCT07053761
Title: A Randomized Controlled Trial of Five - Flavor Sophora Flavescens Enteric - Coated Capsules for Radiation - Induced Proctitis After Pelvic Radiotherapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Shangbin QIN, Doctor, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-206
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Radiation - Induced Proctitis
Keywords: radiation - induced proctitis
MeSH Terms: interventions — Glutamine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Drug: five - flavor sophora flavescens enteric - coated capsules plus glutamine and warm - water sitz baths
- control group (Active Comparator)
  Interventions: Drug: glutamine and warm - water sitz baths

INTERVENTIONS:
Drug: five - flavor sophora flavescens enteric - coated capsules plus glutamine and warm - water sitz baths — Experimental group: If patients have rectal reactions, RTOG radiation - therapy toxicity grades >2, plus FOB (+) or fecal calprotectin Fc>150μg/g, they'll take five - flavor sophora flavescens enteric - coated capsules (4 capsules thrice daily for 8 weeks), plus glutamine and warm - water sitz baths.
  Arms: Experimental group
Drug: glutamine and warm - water sitz baths — If patients have rectal reactions, RTOG radiation - therapy toxicity grades >2, plus FOB (+) or fecal calprotectin Fc>150μg/g, they'll use only glutamine and warm - water sitz baths.
  Arms: control group

SUMMARY:
The goal of this single - center, prospective, randomized controlled study is to assess the therapeutic effects of five - flavor sophora flavescens enteric - coated capsules on radiation - induced proctitis in patients who have undergone pelvic radiotherapy. The main question it aims to answer is:

Does five - flavor sophora flavescens enteric - coated capsules treatment improve radiation - induced proctitis in these patients? Participants with radiation - induced proctitis following pelvic radiotherapy will be randomly allocated to either the trial group (receiving the capsules) or the control group (receiving conventional therapy). Assessments will be conducted to compare outcomes between the two groups.

ELIGIBILITY:
Inclusion Criteria:

Aged 18 - 80 years. Undergoing pelvic radiotherapy with RTOG radiation - toxicity grade ≥2 and FOB (+) or fecal calprotectin Fc>150μg/g.

Absolute neutrophil count >1,500/μL, platelets >100,000/μL; AST <45U/L, ALT <40U/L; creatinine clearance >50ml/min.

Willing to sign consent and participate in required tests and follow - up.

Exclusion Criteria:

Previous pelvic/abdominal radiotherapy. Other severe intestinal diseases (e.g., Crohn's, ulcerative colitis, colorectal cancer).

Contraindications to five - flavor sophora flavescens enteric - coated capsules (e.g., prolonged QTc, hypokalemia, use of QTc - prolonging drugs, heart disease).

Allergy to the capsules or their components. Other therapies for radiation - induced proctitis (e.g., mesalamine, steroids, hyperbaric oxygen, laser therapy) in the past month.

Uncontrolled diseases that may affect the study, such as organ dysfunction, poorly controlled hypertension, coronary heart disease, arrhythmias, cerebrovascular disease, diabetes; myocardial infarction or heart failure in the past 6 months; jaundice due to hepatic insufficiency; AIDS; uncontrolled coagulation disorders.

Psychiatric patients unable to complete the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical remission rate of acute radiation rectal injury | 3 months
  Clinical remission rate of acute radiation rectal injury